CLINICAL TRIAL: NCT05720650
Title: B Vitamin Deficiency and Pregnancy Complications
Status: Withdrawn | Type: Observational
Why Stopped: plans changed
Sponsor: Westlake University (Other)
Collaborators: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Other Study IDs: WestlakeU
Record Dates: First submitted 2022-11-14; First posted 2023-02-09 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2022-11

CONDITIONS: Gestational Hypertension; Preeclampsia
Keywords: B vitamins; pregnancy complications
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; Pregnancy Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — maternal blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case subjects diagnosed with gestational hypertension or preeclampsia: This is a restrospective observational study and there is no intervention.
  Interventions: Other: No intervention
- Control subjects diagnosed without any hypertensive disorders: This is a restrospective observational study and there is no intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This case-control study aims to investigate the association between B vitamins and gestational hypertension or preeclampsia.

DETAILED DESCRIPTION:
In clinical practice, women diagnosed with gestational hypertension or preeclampsia will be asked to participate this study to fill a questionnaire reporting their basic information. Meanwhile, women with matched age and gestation week and without any kinds of hypertensive disorders will also be invited for this study. Participants' blood samples will be analyzed for B vitamin levels at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women aged 18-40 years old

Exclusion Criteria:

* women with Hepatitis B, syphilis, HIV/AIDS and other infectious diseases.
* women with severe physical or mental diseases

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: pregnant women aged 18-45 years old
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
gestational hypertension | seven days after delivery
  Gestational hypertension is diagnosed when blood pressure readings are higher than 140/90 mm Hg in a woman who had normal blood pressure prior to 20 weeks and has no proteinuria (excess protein in the urine).
preeclampsia | seven days after delivery
  Gestational hypertension is diagnosed when blood pressure readings are higher than 140/90 mm Hg in a woman who had normal blood pressure prior to 20 weeks and has positive proteinuria (excess protein in the urine).

CONTACTS AND LOCATIONS:
Overall Officials: Hongjun SHI, PhD, Principal Investigator — Westlake University
Locations (1):
- Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided